CLINICAL TRIAL: NCT01735201
Title: AGN-199201 for the Treatment of Erythema With Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 199201-002
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Rosacea; Erythema
MeSH Terms: conditions — Rosacea; Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- AGN-199201 Dose A Once Daily (Experimental): AGN-199201 Dose A applied once daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Dose A
- AGN-199201 Dose B Once Daily (Experimental): AGN-199201 Dose B applied once daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Dose B
- AGN-199201 Dose C Once Daily (Experimental): AGN-199201 Dose C applied once daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Dose C
- AGN-199201 Vehicle Once Daily (Placebo Comparator): AGN-199201 Vehicle applied once daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Vehicle
- AGN-199201 Dose A Twice Daily (Experimental): AGN-199201 Dose A applied twice daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Dose A
- AGN-199201 Dose B Twice Daily (Experimental): AGN-199201 Dose B applied twice daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Dose B
- AGN-199201 Dose C Twice Daily (Experimental): AGN-199201 Dose C applied twice daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Dose C
- AGN-199201 Vehicle Twice Daily (Placebo Comparator): AGN-199201 Vehicle applied twice daily to the face for 28 days.
  Interventions: Drug: AGN-199201 Vehicle

INTERVENTIONS:
Drug: AGN-199201 Dose A — AGN-199201 Dose A applied once or twice daily to the face for 28 days.
  Arms: AGN-199201 Dose A Once Daily; AGN-199201 Dose A Twice Daily
Drug: AGN-199201 Dose B — AGN-199201 Dose B applied once or twice daily to the face for 28 days.
  Arms: AGN-199201 Dose B Once Daily; AGN-199201 Dose B Twice Daily
Drug: AGN-199201 Dose C — AGN-199201 Dose C applied once or twice daily to the face for 28 days.
  Arms: AGN-199201 Dose C Once Daily; AGN-199201 Dose C Twice Daily
Drug: AGN-199201 Vehicle — AGN-199201 Vehicle applied once or twice daily to the face for 28 days.
  Arms: AGN-199201 Vehicle Once Daily; AGN-199201 Vehicle Twice Daily

SUMMARY:
This study will evaluate the safety and efficacy of 3 doses of AGN-199201 once and twice daily compared to vehicle for the treatment of moderate to severe facial erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Redness of the skin caused by rosacea

Exclusion Criteria:

* ≥3 inflammatory lesions
* Laser light-source or other energy based therapy in the last 6 months
* Any prescription or over the counter product for the treatment of acne or rosacea in the last 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 357 patients were randomized; 1 patient in error. 356 patients were included in the Modified intent-to-treat and Safety populations.
Period: Overall Study
Arm/Group | AGN-199201 Dose A Once Daily | AGN-199201 Dose B Once Daily | AGN-199201 Dose C Once Daily | AGN-199201 Vehicle Once Daily | AGN-199201 Dose A Twice Daily | AGN-199201 Dose B Twice Daily | AGN-199201 Dose C Twice Daily | AGN-199201 Vehicle Twice Daily
Started | 45 | 44 | 44 | 44 | 45 | 45 | 45 | 44
Completed | 42 | 43 | 44 | 42 | 44 | 40 | 42 | 42
Not Completed | 3 | 1 | 0 | 2 | 1 | 5 | 3 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 1 | 3 | 2 | 1
Not completed — Personal Reasons | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Miscellaneous Reasons | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-199201 Dose A Once Daily | AGN-199201 Dose B Once Daily | AGN-199201 Dose C Once Daily | AGN-199201 Vehicle Once Daily | AGN-199201 Dose A Twice Daily | AGN-199201 Dose B Twice Daily | AGN-199201 Dose C Twice Daily | AGN-199201 Vehicle Twice Daily | Total
Number analyzed (Participants) | 45 | 44 | 44 | 44 | 45 | 45 | 45 | 44 | 356
Age, Customized [Number; unit: Participants]
  < 45 years | 14 | 15 | 10 | 14 | 16 | 11 | 16 | 9 | 105
  45-64 years | 30 | 23 | 28 | 24 | 26 | 29 | 27 | 28 | 215
  >= 65 years | 1 | 6 | 6 | 6 | 3 | 5 | 2 | 7 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 33 | 38 | 41 | 34 | 36 | 33 | 285
  Male | 10 | 9 | 11 | 6 | 4 | 11 | 9 | 11 | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 2-Grade Decrease From Baseline on Both Clinician Erythema Assessment (CEA) and Subject Self-Assessment (SSA)
Description: Percentage of participants with at least a 2-grade decrease from Baseline (Improvement) in the CEA score and at least a 2-grade decrease from Baseline (Improvement) in the SSA score were assessed on Day 28 hours 2 to 12. The investigator evaluated the severity of the participant's erythema (redness of the skin) as measured by the CEA using a 5-point scale where 0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness and 4=severe erythema, fiery redness. The participant assessed the severity of their erythema as measured by the SSA using a 5-point scale where 0=clear of unwanted redness; 1=nearly clear of unwanted redness; 2=somewhat more redness than I prefer; 3=more redness than I prefer and 4=completely unacceptable redness.
Time Frame: Baseline, Day 28-hours 2 to 12
Population: Modified intent-to-treat population included all randomized patients who applied study medication during the study, had both CEA and SSA measurements at Baseline and at least 1 post-baseline measurement for both CEA and SSA.
Measure: Number; unit: Percentage of participants
Arm/Group | AGN-199201 Dose A Once Daily | AGN-199201 Dose B Once Daily | AGN-199201 Dose C Once Daily | AGN-199201 Vehicle Once Daily | AGN-199201 Dose A Twice Daily | AGN-199201 Dose B Twice Daily | AGN-199201 Dose C Twice Daily | AGN-199201 Vehicle Twice Daily
Number analyzed (Participants) | 45 | 44 | 44 | 44 | 45 | 45 | 45 | 44
Percentage of participants
  Hour 2 | 13.3 | 20.5 | 22.7 | 6.8 | 8.9 | 17.8 | 15.6 | 6.8
  Hour 4 | 17.8 | 31.8 | 27.3 | 4.5 | 11.1 | 20.0 | 22.2 | 6.8
  Hour 6 | 17.8 | 22.7 | 13.6 | 4.5 | 11.1 | 13.3 | 24.4 | 4.5
  Hour 8 | 15.6 | 20.5 | 20.5 | 4.5 | 8.9 | 20.0 | 20.0 | 2.3
  Hour 10 | 17.8 | 20.5 | 13.6 | 4.5 | 13.3 | 15.6 | 26.7 | 2.3
  Hour 12 | 13.3 | 13.6 | 13.6 | 2.3 | 13.3 | 11.1 | 15.6 | 4.5

2. Secondary Outcome: Percentage of Participants With at Least a 2-Grade Decrease From Baseline on Both CEA and SSA at 0.5 Hour Post-Dose on Day 28
Description: Percentage of participants with at least a 2-grade decrease from Baseline (Improvement) in the CEA score and at least a 2-grade decrease from Baseline (Improvement) in the SSA score were assessed at 0.5 hour post-dose on Day 28. The investigator evaluated the severity of the participant's erythema (redness of the skin) as measured by the CEA using a 5-point scale where 0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness and 4=severe erythema, fiery redness. The participant assessed the severity of their erythema as measured by the SSA using a 5-point scale where 0=clear of unwanted redness; 1=nearly clear of unwanted redness; 2=somewhat more redness than I prefer; 3=more redness than I prefer and 4=completely unacceptable redness.
Time Frame: Baseline, Day 28-hour 0.5
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AGN-199201 Dose A Once Daily | AGN-199201 Dose B Once Daily | AGN-199201 Dose C Once Daily | AGN-199201 Vehicle Once Daily | AGN-199201 Dose A Twice Daily | AGN-199201 Dose B Twice Daily | AGN-199201 Dose C Twice Daily | AGN-199201 Vehicle Twice Daily
Number analyzed (Participants) | 45 | 44 | 44 | 44 | 45 | 45 | 45 | 44
Percentage of participants | 6.7 | 11.4 | 6.8 | 4.5 | 6.7 | 6.7 | 6.7 | 2.3

3. Secondary Outcome: Percentage of Participants With at Least a 2-Grade Decrease From Baseline on Both CEA and SSA at 1 Hour Post-Dose on Day 28
Description: Percentage of participants with at least a 2-grade decrease from Baseline (Improvement) in the CEA score and at least a 2-grade decrease from Baseline (Improvement) in the SSA score were assessed at 1 hour post-dose on Day 28. The investigator evaluated the severity of the participant's erythema (redness of the skin) as measured by the CEA using a 5-point scale where 0=clear skin with no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness and 4=severe erythema, fiery redness. The participant assessed the severity of their erythema as measured by the SSA using a 5-point scale where 0=clear of unwanted redness; 1=nearly clear of unwanted redness; 2=somewhat more redness than I prefer; 3=more redness than I prefer and 4=completely unacceptable redness.
Time Frame: Baseline, Day 28-hour 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AGN-199201 Dose A Once Daily | AGN-199201 Dose B Once Daily | AGN-199201 Dose C Once Daily | AGN-199201 Vehicle Once Daily | AGN-199201 Dose A Twice Daily | AGN-199201 Dose B Twice Daily | AGN-199201 Dose C Twice Daily | AGN-199201 Vehicle Twice Daily
Number analyzed (Participants) | 45 | 44 | 44 | 44 | 45 | 45 | 45 | 44
Percentage of participants | 11.1 | 13.6 | 18.2 | 2.3 | 6.7 | 11.1 | 8.9 | 2.3

ADVERSE EVENTS:
Arm/Group | AGN-199201 Dose A Once Daily | AGN-199201 Dose B Once Daily | AGN-199201 Dose C Once Daily | AGN-199201 Vehicle Once Daily | AGN-199201 Dose A Twice Daily | AGN-199201 Dose B Twice Daily | AGN-199201 Dose C Twice Daily | AGN-199201 Vehicle Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/44 | 0/44 | 1/44 | 0/45 | 1/45 | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 5/45 | 5/44 | 1/44 | 1/44 | 2/45 | 6/45 | 7/45 | 6/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-199201 Dose A Once Daily (N=45) | AGN-199201 Dose B Once Daily (N=44) | AGN-199201 Dose C Once Daily (N=44) | AGN-199201 Vehicle Once Daily (N=44) | AGN-199201 Dose A Twice Daily (N=45) | AGN-199201 Dose B Twice Daily (N=45) | AGN-199201 Dose C Twice Daily (N=45) | AGN-199201 Vehicle Twice Daily (N=44)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Event not related to study treatment.
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Event not related to study treatment.
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Event not related to study treatment.
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Event not related to study treatment.
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Event not related to study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-199201 Dose A Once Daily (N=45) | AGN-199201 Dose B Once Daily (N=44) | AGN-199201 Dose C Once Daily (N=44) | AGN-199201 Vehicle Once Daily (N=44) | AGN-199201 Dose A Twice Daily (N=45) | AGN-199201 Dose B Twice Daily (N=45) | AGN-199201 Dose C Twice Daily (N=45) | AGN-199201 Vehicle Twice Daily (N=44)
Application site dermatitis (General disorders) | 0 | 3 | 0 | 0 | 1 | 3 | 2 | 0
Application site acne (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 3
Headache (Nervous system disorders) | 4 | 1 | 0 | 1 | 1 | 3 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.